CLINICAL TRIAL: NCT01518985
Title: A Phase 1, Placebo-Controlled Trial to Evaluate the Impact of Intravenous (IV) Bendavia™ (MTP-131) on Endothelial Reactivity Dysfunction Induced by Cigarette Smoking
Brief Title: The Impact of Intravenous Bendavia™ on Endothelial Reactivity Dysfunction in Cigarette Smoking
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SPIRI-120
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Intravenous infusion of saline (0.9%) for 4 hours with smoking of one unfiltered cigarette at 30 minutes post-study-drug administration start
  Interventions: Drug: Sterile saline (0.9%); Other: Cigarette smoking
- Bendavia (Experimental): Intravenous infusion of Bendavia (0.25mg/kg/hr) for 4 hours with smoking of one unfiltered cigarette at 30 minutes post-study-drug administration start
  Interventions: Drug: Bendavia; Other: Cigarette smoking

INTERVENTIONS:
Drug: Bendavia — Bendavia for infusion Intravenous infusion (0.25mg/kg/hr) for 4 hours
  Arms: Bendavia
Drug: Sterile saline (0.9%) — Sterile saline for infusion (0.9%) Intravenous infusion for 4 hours
  Arms: Placebo
Other: Cigarette smoking — One unfiltered cigarette will be smoked at approximately 30 minutes post-study-drug administration start.

SUMMARY:
This will be a phase 1 randomized, double-blind, 2-period, 2-sequence crossover trial enrolling 6 healthy volunteers to assess the impact of IV-administered Bendavia on the endothelial dysfunction induced by a single cigarette.

ELIGIBILITY:
Inclusion Criteria:

- Healthy adult male smokers between 18 and 65 years of age with signed informed consent

Exclusion Criteria:

* Serum sodium level below the lower limit of sites' clinical laboratory normal range at screening, D-1 and 6
* Cholesterol level ≥ 240 mg/dL
* Hypertension (blood pressure SBP > 140, DBP > 90 mmHg)
* Body mass index < 18 or > 32 kg/m2,
* Creatinine clearance calculated by the Cockcroft and Gault method calculated to be < 90 mL/min,
* Additional laboratory abnormalities determined as clinically significant by the Principal Investigator at laboratory screening
* Clinically significant abnormalities on physical examination,
* History or evidence of renal, hepatic, pulmonary (including chronic asthma), endocrine (e.g., diabetes), central nervous, or gastrointestinal (including an ulcer) system dysfunction,
* History of seizures or history of epilepsy,
* History of serious (Principal Investigator judgment) mental illness,
* Receipt of investigational medicinal product within 30 days prior to the planned date of study drug administration,
* Positive serology for human immunodeficiency virus type 1 or 2, or hepatitis B surface antigen,
* Fever > 37.5°C at the time of planned dosing,
* Suspicion, or recent history, of alcohol or substance abuse,
* Donated blood or blood products within the past 30 days,
* Employee or family member of the investigational site,
* Subjects who are either unwilling to agree to refrain from use or found to be using Nicotine (or nicotine products) including cigarettes from 12 hours prior to start of each study drug infusion through to the completion of endothelial function testing, Alcohol, Caffeine, Xanthine-containing food or beverages and over-the-counter medications with the exception of Tylenol from 24 hours prior to dosing and throughout the confinement periods, Supplementary antioxidant vitamins from 7 days prior to dosing and throughout the confinement periods, Prescription medications from 14 days prior to and 7 days post treatment
* Subjects having previous exposure to Bendavia.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Analysis of variance (ANOVA) between group mean endothelial function (EndoPAT Index) following smoking a single cigarette with and without Bendavia | Baseline, +30, +60, +90 minutes post-study-drug administration start
  Endothelial function will be determined using EndoPAT 2000 (Itamar Medical Ltd) prior to and after smoking of one unfiltered cigarette and prior to and after initiation of study drug. Group comparison of endothelial function (EndoPAT Index) between placebo and active study drug within a subject will be performed.
  EndoPAT quantifies the endothelium-mediated changes in vascular tone. A post-occlusion to pre-occlusion ratio is calculated providing the EndoPAT index.

SECONDARY OUTCOMES:
Anova between group mean inflammatory laboratory marker (hs-CRP; mg/L) after smoking one cigarette with and without Bendavia | Baseline to 24 hours post-study-drug administration
  hs-CRP will be evaluated prior to and after smoking of one unfiltered cigarette and prior to and after initiation of study drug. Group comparison of hs-CRP levels between placebo and active study drug within a subject will be performed.
ANOVA between group means of urinary 8-isoprostane (ng/mg of creatinine) after smoking one cigarette with and without Bendavia | Baseline to 48 hours post-study-drug administration
  8-isoprostane will be measured prior to and after smoking of one unfiltered cigarette and prior to and after initiation of study drug. Group comparison of laboratory results between placebo and active study drug within a subject will be performed.
Number adverse events with and without Bendavia | Baseline to Study Day 10
  Adverse events will be tabulated by treatment group. No statistical analysis will be preformed.
Assessment of Bendavia exposure measured by area Under the Curve (AUC; ng*hr/mL) | Baseline to 48 hours post-study-drug administration
  Bendavia levels will be measured and pharmacokinetic parameters reported.
ANOVA between group means of urinary 8-hydroxy-2'-deoxyguanosine (pg/mL) after smoking one cigarette with and without Bendavia | Baseline to 48 hours post-study-drug administration
  8-hydroxy-2'-deoxyguanosine will be measured prior to and after smoking of one unfiltered cigarette and prior to and after initiation of study drug. Group comparison of laboratory results between placebo and active study drug within a subject will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C Lasseter, MD, Principal Investigator — Clinical Pharmacology of Miami; Richard Straube, MD, Study Director — Stealth Peptides
Locations (1):
- Clinical Pharmaology of Miami, Miami, Florida, United States